CLINICAL TRIAL: NCT00687401
Title: A Multi-center, Open Label Trial Evaluating the Efficacy , SAfety and the Impact on QUAlity of Life of Infliximab TherapY in Patients With Moderate-to-severe Psoriasis Not Responding to Standard or Biologic Therapy
Brief Title: A Study to Evaluate Infliximab in Subjects With Moderate-to-Severe Psoriasis Not Responding to Standard or Biologic Therapy (Study P04612)
Acronym: ESAQUALITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04612
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2010-12-24 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Infliximab 5 mg/kg (Experimental): Infliximab 5 mg/kg of body weight administered as an infusion at Weeks 0, 2, 6, and 14.
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — Infliximab 5 mg/kg of body weight administered as an infusion at Weeks 0, 2, 6 (induction phase), and 14 (maintenance phase).
  Other Names: Remicade, SCH 215596

SUMMARY:
Subjects with moderate-to-severe chronic psoriasis not responding to standard or biologic therapy will be eligible to enroll in this study. Subjects will receive infliximab infusions (5 mg/kg of body weight) at Weeks 0, 2, 6, and 14 followed by a 12-week follow-up period. The efficacy of infliximab will be evaluated by the Psoriasis Area and Severity Index (PASI).

ELIGIBILITY:
Inclusion Criteria:

* >=18 to 75 years of age, of either gender, and of any race.
* Psoriasis covering at least 10% of total body surface area (BSA) and PASI >=12 at Screening and Baseline.
* Diagnosis of moderate-to-severe psoriasis at least 6 months prior the screening.
* Eligible to infliximab who have failed at least 1 of the following: corticosteroids, methotrexate (MTX), systemic retinoids, cyclosporine, psoralen-ultraviolet A (PUVA), ultraviolet B (UVB) phototherapy, and/or biologics (etanercept or efalizumab).
* Eligible according to tuberculosis (TB) eligibility assessment, screening and early detection of reactivation rules.
* Chest x-ray within 3 months prior to Screening with no evidence of malignancy, infection, or fibrosis.
* Screening and Baseline tests (complete blood count [CBC], blood chemistry, and urinalysis) must be within protocol-specified parameters.
* Free of significant disease that could interfere with study evaluations.
* Willing to give written informed consent and able to adhere to protocol visits and procedures.
* Women of childbearing potential and all men must be using adequate birth control and must continue to do so for 6 months after receiving the last dose of study medication.
* Females of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline.

Exclusion Criteria:

* Standard concomitant psoriasis therapies.
* Active or latent TB.
* History of chronic infectious disease, opportunistic infection, or serious infection within 2 months of enrollment.
* History of lymphoproliferative disease.
* Malignancy in past 5 years (except treated basal cell carcinoma [BCC]).
* Treatment with tumor necrosis factor (TNF) antagonists within previous 6 weeks.
* Current drug-induced psoriasis.
* Females who are pregnant or nursing and females and males who are planning pregnancy within 6 months from the last infusion of infliximab.
* Previously treated with infliximab.
* Concomitant diagnosis of congestive heart failure (CHF) including medically-controlled asymptomatic subjects.
* History of chronic or recurrent infectious disease.
* Have or have had a serious infection or have been hospitalized or received intravenous antibiotics for an infection during the 2 months prior to Screening.
* Have or have had an opportunistic infection within 6 months prior to Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2006-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Infliximab 5 mg/kg: Infliximab 5 mg/kg of body weight administered as an infusion at Weeks 0, 2, 6 (induction phase), and 14 (maintenance phase).
Period: Overall Study
Arm/Group | Infliximab 5 mg/kg
Started | 159 (215 participants enrolled in the study, of which 56 failed screening and did not receive study drug.)
Completed | 129
Not Completed | 30
Not completed — Protocol Violation | 7
Not completed — Adverse Event | 6
Not completed — Lack of Efficacy | 6
Not completed — Withdrawal by Subject | 4
Not completed — Did not return for visit | 3
Not completed — For reasons different from those above | 4

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.15 (12.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 119

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieve a Greater Than or Equal to 75% Improvement in Psoriasis Area and Severity Index (PASI) Score
Description: PASI 75 response is defined as participants who achieved at least a
  75% improvement in PASI score from Baseline to Week 10. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their responses to therapy. The PASI produces a numeric score that can range from 0 to 72 (the higher the number, the worse the disease).
Time Frame: 10 weeks
Population: Intent to Treat Population (ITT): 159 participants out of the 215 enrolled patients who received at least one dose of the study drug.
  Per Protocol Population (PP): 138 participants not withdrawn from the study due to major protocol violation and who have received the three infusions of the study drug planned by the protocol.
Measure: Number; unit: Participants
Groups:
- Intent to Treat Population; Per Protocol Population: Infliximab 5 mg/kg of body weight administered as an infusion at Weeks 0, 2, 6 (induction phase), and 14 (maintenance phase).
Arm/Group | Intent to Treat Population | Per Protocol Population
Number analyzed (Participants) | 159 | 138
Participants | 111 | 111

ADVERSE EVENTS:
Arm/Group | Infliximab 5 mg/kg
Serious Adverse Events (participants affected / at risk) | 2/159
Other Adverse Events (participants affected / at risk) | 16/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab 5 mg/kg (N=159)
pneumonia legionella (Infections and infestations) | 1 (1)
erythema (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab 5 mg/kg (N=159)
pyrexia (General disorders) | 9 (10)
arthralgia (Musculoskeletal and connective tissue disorders) | 8 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No specific time period restrictions. If the parties disagree concerning the accuracy and appropriateness of the data analysis and presentation, and/or confidentiality of information, the Sponsor and the Investigator will make good faith efforts to resolve any issues or disagreement.